CLINICAL TRIAL: NCT06149962
Title: Comparison Between Functional Outcomes of Flexor Tendon Repair Under Wide Awake Local Anesthesia no Tourniquet and Brachial Plexus Block
Brief Title: Comparison Between Functional Outcomes of Flexor Tendon Repair Under WALANT and Brachial Plexus Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Omar Mohamed Hussein, Resident-plastic department-sohag hospital university, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: soh_med_23_06_07ms
Record Dates: First submitted 2023-08-06; First posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Flexor Tendon Rupture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WALANT (Active Comparator): Flexor Tendon Repair under Wide-Awake Local Anesthesia No Tourniquet
  Interventions: Procedure: FLEXOR TENDON REPAIR
- BRACHIAL BLOCK (Active Comparator): Flexor Tendon Repair under Brachial Plexus Block
  Interventions: Procedure: FLEXOR TENDON REPAIR

INTERVENTIONS:
Procedure: FLEXOR TENDON REPAIR — we will repair tendon of FDP only using 6 strand technique using PDS 4/0 core suture - prolene 6/0 running suture under WALANT technique and brachial plexus block.

SUMMARY:
Although outcomes after flexor tendon repair have reportedly improved with modern treatment, complications are common. Early passive and active motion protocols have improved outcomes of flexor tendon repairs. One potential complication of early motion occurs when the forces produced by this motion exceed the strength of the repair, which leads to gap formation and inhibits healing. Wide Awake Local Anesthesia No Tournique (WALANT) is a new anesthesia technique that has gained popularity among plastic surgeons. It was developed by Dr. Lalonde in Canada, and it involves the use of Lidocaine and adrenaline in the surgical site to control bleeding without the need for a tourniquet. Peripheral nerve blocks are overall safe when performed correctly, there are rare but serious risks associated with them. Risks include block failure, bleeding, infection, damage to surrounding structures, permanent nerve injury, and intravascular uptake of local anesthetic resulting in systemic toxicity.

DETAILED DESCRIPTION:
WALANT can be applied in both elective and emergency surgeries and is commonly used for procedures involving the hand, wrist, and fingers, such as root tunnels syndromes, trigger finger, and fractures. However, it has some limitations and contraindications, including patients with coagulopathy or on anticoagulant therapy, those with allergies to any of the anesthesia components, or patients with a history of psychiatric disorders or aggressive behavior. Infraclavicular brachial plexus block (ICBPB) is widely used for anesthesia or analgesia during surgery on the hand and forearm. Today, it is most frequently performed using a sagittal ultrasound scan at the lateral infraclavicular fossa (LICF), where the local anesthetic is injected deep to the pectoral muscles. Peripheral nerve blocks are overall safe when performed correctly, there are rare but serious risks associated with them. Risks include block failure, bleeding, infection, damage to surrounding structures, permanent nerve injury, and intravascular uptake of local anesthetic resulting in systemic toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Cooperative patients .
* age between 16-60 years.
* Acute flexor tendon injuries of the hand in both genders in medial four fingers.
* Sharp mechanism of injury.
* Single level injury zone 2.

Exclusion Criteria:

* Associated fractures close to the tendon injury.

  * Vascular injury requiring revascularization
  * Multiple level injury
  * Combined flexor and extensor laceration
  * Insufficient skin and soft tissue coverage
  * Tendon substance loss
  * Patients with coagulopathy or on anticoagulant therapy
  * Patients with allergies to any of the anesthesia components

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-07-10 (Estimated); Study Completion 2024-07-10 (Estimated)

PRIMARY OUTCOMES:
Quick Disabilities of the Arm, Shoulder, and Hand | 6 months
  Quick Disabilities of the Arm, Shoulder, and Hand using (DASH) scores

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed G ABDELMAGEED, A.PROF, Study Chair — SOHAG U
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
YES

REFERENCES:
- [Background] Dy CJ, Hernandez-Soria A, Ma Y, Roberts TR, Daluiski A. Complications after flexor tendon repair: a systematic review and meta-analysis. J Hand Surg Am. 2012 Mar;37(3):543-551.e1. doi: 10.1016/j.jhsa.2011.11.006. Epub 2012 Feb 6. PMID 22317947
- [Background] Lalonde D. How the wide awake approach is changing hand surgery and hand therapy: inaugural AAHS sponsored lecture at the ASHT meeting, San Diego, 2012. J Hand Ther. 2013 Apr-Jun;26(2):175-8. doi: 10.1016/j.jht.2012.12.002. Epub 2013 Jan 5. No abstract available. PMID 23294825
- [Background] Pollard R, Higham H, Quinlan J, Webster R, Lie J, Sivasubramaniam S. Nerve block site marking. Anaesthesia. 2019 Jan;74(1):123-124. doi: 10.1111/anae.14527. No abstract available. PMID 30511750
- [Background] Sotthisopha T, Elgueta MF, Samerchua A, Leurcharusmee P, Tiyaprasertkul W, Gordon A, Finlayson RJ, Tran DQ. Minimum Effective Volume of Lidocaine for Ultrasound-Guided Costoclavicular Block. Reg Anesth Pain Med. 2017 Sep/Oct;42(5):571-574. doi: 10.1097/AAP.0000000000000629. PMID 28723837